CLINICAL TRIAL: NCT06195254
Title: A Retrospective Clinical Study of Stereotactic Body Radiotherapy Combined With PD-1 Blockers for Locally Advanced or Locally Recurrent Pancreatic Carcinoma.
Brief Title: Stereotactic Body Radiotherapy Combined With PD-1 Blockers for Locally Advanced or Locally Recurrent Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: preSPARK-1
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2020-12

CONDITIONS: Stereotactic Body Radiotherapy; PD-1 Inhibitors; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SBRT+PD-1 blockers: pembrolizumab (200 mg every 3 weeks), carelizumab (200 mg every 3 weeks), tislelizumab (200 mg every 3 weeks), sintilimab (200 mg every 3 weeks), zimberelimab (240 mg every 3 weeks) until the tumor progressed or the side effects became intolerable.
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: PD-1 blocking antibody

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — All the patients first received SBRT with the dose of 25Gy up to 50Gy in five fractions.
Drug: PD-1 blocking antibody — All the patients first received SBRT with the dose of 25Gy up to 50Gy in five fractions and then received the treatment of PD-1 blockers including pembrolizumab (200 mg every 3 weeks), carelizumab (200 mg every 3 weeks), tislelizumab (200 mg every 3 weeks), sintilimab (200 mg every 3 weeks), zimberelimab (240 mg every 3 weeks) until the tumor progressed or the side effects became intolerable.

SUMMARY:
The goal of this observational study is to investigate the efficacy and safety of stereotactic body radiotherapy combined with PD-1 blockers for LAPC and LRPC. The patients, diagnosed with locally advanced pancreatic cancer (LAPC) or locally recurrent pancreatic cancer (LRPC). LRPC or LAPC, undergoing SABT and PD-1 blockers in our hospital from December 2020 to April 2023 were reviewed consecutively. All patients provided written informed consent before treatment. The study was conducted in accordance with the Declaration of Helsinki, and it was approved by the Institutional Ethics Committee of Peking University Third Hospital.

DETAILED DESCRIPTION:
The goal of this observational study is to investigate the efficacy and safety of stereotactic body radiotherapy (SBRT) combined with PD-1 blockers for LAPC and LRPC. The patients, diagnosed with locally advanced pancreatic cancer (LAPC) or locally recurrent pancreatic cancer (LRPC). LRPC or LAPC, undergoing SBRT and PD-1 blockers in our hospital from December 2020 to April 2023 were reviewed consecutively. The schedule of SBRT is 25 to 50 Gy in 5 fractions and the PD-1 blockers are monoclonal antibodies targeted to PD-1 molecules on the T lymphocytes.

All patients provided written informed consent before treatment. The study was conducted in accordance with the Declaration of Helsinki, and it was approved by the Institutional Ethics Committee of Peking University Third Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. LRPC confirmed by pathologic or imaging diagnosis and LAPC confirmed by pathology;
2. disease size ≥1 cm;
3. KPS≥70;
4. adequate hematological reserves, hepatic function, renal function and heart function;
5. expected survival > 3 months.

Exclusion Criteria:

1. unconfirmed mass;
2. The upper abdomen was previously treated with radiotherapy;
3. the patients previously underwent immunotherapy of PD-1 or PD-L1 monoclonal antibody;
4. a history of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency or other immune-related conditions requiring long-term oral hormone therapy;
5. patients with active infectious disease, trauma and severe wounds;
6. patients with any mental disorder;
7. patients with other somatic comorbidities of clinical concern;
8. pregnancy and lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients, diagnosed with LRPC or LAPC, undergoing SABT and PD-1 blockers in our hospital from December 2020 to April 2023 were reviewed consecutively. All patients provided written informed consent before treatment. The study was conducted in accordance with the Declaration of Helsinki, and it was approved by the Institutional Ethics Committee of Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 12 months
  PFS was defined as the time from SBRT to disease progression

SECONDARY OUTCOMES:
local progression-free survival (LPFS) | 12 months
  LPFS was defined as the time from SBRT to local progression.
Overall survival (OS) | 18 months
  OS was defined as the time from SBRT to death from any cause.
Adverse Events (AEs) | 18 months
  All kinds of side effects.
Pain relief rate (PRR） | 18 months
  The numeric rating scale (NRS) was used to evaluate the pain levels before and after treatment and the pain relief rate was calculated from the patients achieving pain The numeric rating scale (NRS) was used to evaluate the pain levels before and after treatment and the pain relief rate was calculated from the patients achieving pain The numeric rating scale (NRS) was used to evaluate the pain levels before and after treatment and the pain relief rate was calculated from the patients achieving pain relief after SBRT.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Junjie Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Allways.
Access Criteria: The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.